CLINICAL TRIAL: NCT04722471
Title: Progesterone Levels and Clinical Outcomes Using a Single Pessary of 400 mg of Vaginal Progesterone in Substitutive Cycles for Embryo Transfer.
Acronym: CycloCT
Status: Completed | Type: Observational
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Joaquín Llácer, Principal Investigator, Instituto Bernabeu
Other Study IDs: IB-1201
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Luteal Phase Defect
Keywords: Frozen embryo transfer; endometrial preparation; artificial cycle; progesterone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 400 mg: Treatments where 400 mg tablet presentation of micronized vaginal progesterone was used, the protocol being one vaginal tablet twice a day.
  Interventions: Drug: Vaginally administered progesterone
- 200 mg: Treatments where 200 mg tablet presentation of micronized vaginal progesterone was used, the protocol being two vaginal tablets twice a day.
  Interventions: Drug: Vaginally administered progesterone

INTERVENTIONS:
Drug: Vaginally administered progesterone — The artificial endometrial preparation for an embryo transfer with the use of 400 mg vaginal tablet (one tablet twice a day) or 200 mg (two tablets twice a day)

SUMMARY:
This study aims to compare the efficacy, in terms of progesterone levels and clinical outcomes, of two different presentations of micronized vaginal progesterone (400 mg vs. 200 mg) used in endometrial preparation in artificial cycle (AC) for embryo transfer.

This is a non-inferiority, retrospective case-control study, with at least 200 cycles analyzed (at least 100 per arm) and the primary outcome is the serum progesterone level on the day of the embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary infertility undergoing endometrial preparation for an embryo transfer using standard doses of oral or transdermal estrogens.
* Age between 18 and 50 years.
* Normal uterine cavity verified by imaging techniques.
* Serum progesterone documented on the day of embryo transfer.

Exclusion Criteria:

* Patients with a history of endometritis.
* Patients diagnosed with Asherman's syndrome.
* Patients with a different supplementation regimen or doses than those of the study groups.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population will be selected among those patients who have undergone embryo transfer treatment with endometrial preparation in a artificial cycle at the Instituto Bernabeu.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Serum progesterone level | On the day of embryo transfer

SECONDARY OUTCOMES:
Need for additional progesterone supplementation | assessed on the day of the embryo transfer
Clinical results (ongoing pregnancy and miscarriage rate) | assessed on the day of the pregnancy test and during the pregnancy evolution

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Llácer, MD PhD, Principal Investigator — Instituto Bernabeu
Locations (1):
- Instituto Bernabeu, Alicante, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
The information collected in the study will always be treated as grouped data and never as individual or personal data, thus maintaining anonymity and confidentiality.

REFERENCES:
- [Result] Labarta E, Mariani G, Holtmann N, Celada P, Remohi J, Bosch E. Low serum progesterone on the day of embryo transfer is associated with a diminished ongoing pregnancy rate in oocyte donation cycles after artificial endometrial preparation: a prospective study. Hum Reprod. 2017 Dec 1;32(12):2437-2442. doi: 10.1093/humrep/dex316. PMID 29040638
- [Result] Labarta E, Mariani G, Paolelli S, Rodriguez-Varela C, Vidal C, Giles J, Bellver J, Cruz F, Marzal A, Celada P, Olmo I, Alama P, Remohi J, Bosch E. Impact of low serum progesterone levels on the day of embryo transfer on pregnancy outcome: a prospective cohort study in artificial cycles with vaginal progesterone. Hum Reprod. 2021 Feb 18;36(3):683-692. doi: 10.1093/humrep/deaa322. PMID 33340402